CLINICAL TRIAL: NCT05376579
Title: Impact of Mayzent (Siponimod) on Active Secondary Progressive Multiple Sclerosis Patients in a Long-term Non-interventional Study in Italy
Brief Title: Impact of Mayzent on aSPMS Patients in a Long-term NIS in Italy
Acronym: ITASIA
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312AIT04
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Active Secondary Progressive Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis; aSPMS; NIS; Italy; Mayzent; siponimod
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — siponimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- siponimod: patients treated with siponimod
  Interventions: Other: siponimod

INTERVENTIONS:
Other: siponimod — Prospective observational cohort study. There is no treatment allocation. Patients will be invited to participate in the study after the independent decision by physician and patient to start siponimod treatment as routine clinical care.
  Other Names: mayzent

SUMMARY:
This is an observational, multicenter, single-arm, prospective study conducted in Italy

DETAILED DESCRIPTION:
Primary data will be collected over a period of three years. Medical history of participants will be collected including EDSS, MRI outcomes, relapses and previous medication to allow the estimation of the effects of siponimod treatment on an individual basis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent: patient must provide written informed consent before any study assessment is performed.
2. Male/female participants aged between 18 and 60.
3. Documented diagnosis of active SPMS.
4. Siponimod treatment as routine medical care: patients newly treated with siponimod (starting not more than 7 days before baseline visit), for whom the decision to start treatment has already been taken independently of study inclusion based on clinical practice and according to SmPC and AIFA criteria, and who successfully qualified for treatment with siponimod (i.e. passed the screening procedure mandated by the SmPC and Risk Management Plan (RMP) for this treatment, including genotyping for CYP2C9 to determine CYP2C9 metaboliser status).

Exclusion Criteria:

1. Patients treated outside the approved siponimod label or with any controindication indicated in the SmPC.
2. Pregnant or lactating women.
3. Patients with any clinical condition that may interfere with the subject's ability to cooperate and comply with the study procedures based on the investigator's judgement.
4. Current participation in an interventional trial.
5. Treatment with siponimod prior to inclusion in this study (siponimod can be started not more than 7 days before baseline visit).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients in Italy with active SPMS treated with siponimod as per label and local clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with six-month CDP during 36 months of treatment | 36 months
  Confirmed disability progression (CDP) is defined as a ≥1.0-point worsening of Expanded Disability Status Scale (EDSS) score from ≤5.0 baseline or a 0.5-point worsening from >5.0 baseline for at least 6 months OR a ≥4.0-point confirmed cognitive worsening (CCW) from baseline of Symbol Digit Modalities Test (SDMT) for at least 6 months.

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) | Month 12, month 24 and month 36
  ARR is the number of relapses during the period / person-years of subject Person-years for subject = period (in days) / 365.25
Number of new/newly enlarging T2 [neT2] and Gd+T1 lesions | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  Number of new/newly enlarging T2-hyperintense lesions and number of new 1 gadolinium-enhancing (Gd+) lesions is collected
Expanded Disability Status Scale scores | Month 12, month 24 and month 36
  Expanded Disability Status Scale (EDSS) score is composed of the overall impression and individual scores of the following functional systems: cognition, mood, fatigue, vision, brain stem, upper extremities, lower extremities, bladder-intestinal function, sexuality. Scores are on a scale of 0 (healthy) to 10 (death from MS) with 0.5 unit increments
Expanded Disability Status Scale trend | Month 12, month 24 and month 36
  EDSS trend is measured by differentiating patients who stabilize from those who experience an increase of EDSS score (increment of ≥1 or ≥0.5 point if baseline EDSS was ≤5.0 or ˃5.0, respectively). Moreover, patients with progression will be categorized as patients with continuous disability accrual (CDA) or one-step worsening (OneS-wors), defined as:
  * OneS-wors: the occurrence of one single episode of confirmed EDSS deterioration.
  * CDA: occurrence of at least two episodes of OneS-wors associated with continuous disability progression between at least two time points.
Proportion of patients with No Evidence of Disease Activity (NEDA)-3 | Month 12, month 24 and month 36
  NEDA-3 is defined as no Confirmed disability progression (CDP), no confirmed relapse and absence of T1 gadolinium-enhancing (Gd+) lesions.
UK Neurological Disability Scale (UKNDS) | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The UKNDS is a questionnaire for recording impairments in MS from the patient's perspective and considers 12 functional systems: perception and thinking, mood, vision, speech and communication, swallowing, arm and hand function, walking ability, bladder function, bowel function, fatigue, sexuality, pain, cramps and others. Answering the questions results in a score of 0 (no disability) to 60 (maximum disability). This questionnaire will be completed by the patients during site visits.
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The FSMC is a patient questionnaire for the clarification of cognitive and motor fatigue, a typical symptom of MS (Penner et al., 2009), and considers a cognitive, motor and total score. Score ranges from 200 to 100, the greater the score the greater the impairment caused by fatigue.
Hospital Anxiety and Depression Scale (HADS) | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The HADS has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
  Calculations of scores: each of the 14 items is rated on a 4-point scale ('Yes, definitely', 'Yes, sometimes', 'No, not much' and 'No, not at all'). All items except 7 and 10 are scored as 'Yes, definitely' = 3 to 'No, not at all' = 0. Items 7 and 10 are scored as 'Yes, definitely' = 0 to 'No, not at all' = 3. The HADS consists of two sub-scores: the HAD-A for anxiety and HAD-D for depression; each sub-score ranges from 0 to 21 points; scores ≥11 indicate the presence of anxious or depressive disorders; scores between 8-10 points are borderline abnormal, and scores of ≤7 indicate that the disorder is not present.
Symbol Digit Modality test (SDMT) | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The SDMT is a sensitive and specific test to investigate attention, concentration and information processing speed, which are typically impaired in cognitively impaired MS patients.
  Nine numbers are shown paired with 9 corresponding individual symbols. Below this are further lines with symbols and empty boxes. The patients must assign the correct numbers to the symbols as quickly as possible. The number of correctly assigned numbers within 90 seconds gives the test score. The total duration of the test is about 5 minutes and scores range between 0 and 110 where higher scores indicate better result.
  A deterioration of the SDMT score by ≥4 points is considered clinically relevant
Clinical Global Impression (CGI) | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The CGI scale represents a short, independent assessment by the treating physician of the overall condition of the patient.
  It incorporates patient history, psychosocial circumstances, symptoms, behavior and the influence of symptoms on the patient's functional ability. The CGI consists of three different global measures and all three will be evaluated: Severity of illness (CGI-S) ranges from 0 to 7, Global Improvement (CGI-I) ranges from 0 to 7 and Efficacy index (CGI-E) ranges from 0 to 16. A higher score means a severe impact on the disease.
MS activity status (MS-AS) - number of relapse | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  Number of relapse, number of relapse that affects the daily activities, number of relapse that required an hospitalization and number of treated relapse to be collected
MS activity status (MS-AS) - Number of patients with presence of symptoms | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  Number of patients with presence of symptoms to be collected
T25-foot-walk | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The T25-FW is an objective and quantitative test of the lower extremities. The time in seconds it takes a patient to walk a distance of 25 feet (7.62 m) is measured. The patient should walk as quickly and safely as possible. This test is performed twice in a row and the mean value of the time required is documented in seconds. An improvement or deterioration of 20% is considered a significant change
9-Hole peg test | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  This test examines manual dexterity. Patients must individually remove nine pegs from a flat dish with one hand and insert them into corresponding holes in a test board. The pegs are then placed back into the dish with the same hand. Two rounds are performed per hand and the average value of the time required is documented in seconds
EQ-5D: EuroQol five-dimensional | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The EQ-5D is a generic multidimensional measurement tool for describing health-related quality of life (EuroQol, 1999). The five domains of mobility, self-care ability, daily activities, pain/discomfort and anxiety/depression are considered. For each of the dimensions, the most appropriate answer from three given possibilities is selected (1=no problem, 2=moderate problem, 3=large problem). In addition, the patient marks the current state of health on a scale from 0 (worst conceivable state of health) to 100 (best conceivable state of health).
TSQM-9: Treatment Satisfaction Questionnaire for Medication | Baseline, month 3, month 6, month 12, month 18, month 24, month 30 and month 36
  The TSQM-9 is a questionnaire to assess patient satisfaction with siponimod treatment. The TSQM-9 is a sound and valid measure of the major dimensions of patients' satisfaction with medication and also a good predictor of adherence across different types of medication and patient population.
  Effectiveness, side effects, simplicity and overall satisfaction are all rated between 0 and 100. Higher values mean a worse condition. Responses to items are summed and transformed so that higher scores indicate greater satisfaction. Specifically, TSQM-9 scale scores are computed by adding the items loading on each domain. The lowest possible score is subtracted from the composite score and divided by the greatest possible score range. This provides a transformed score between 0 and 1 that is then multiplied by 100. If more than one item is missing from a subscale of the TSQM-9 for a particular patient, this subscale should be considered invalid for that respondent.
Exposure adjusted proportion of patients with adverse event (AE) or serious adverse event (SAE) per 100 subject-years | Up to 36 months
  Exposure adjusted proportion of patients with adverse event (AE) or serious adverse event (SAE) per 100 subject-years to be collected
Discontinuation rates due to AE or other reasons | Up to 36 months
  Discontinuation rates due to AE or other reasons to be collected
Proportion of patient who required FDO when starting siponimod and the reason why | Baseline
  Proportion of patient who required first dose observation (FDO) when starting siponimod and the reason why

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Italy (21):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Como, CO
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara

IPD SHARING:
Plan to Share IPD: No